CLINICAL TRIAL: NCT03581903
Title: A Phase I Study in Healthy Adults to Assess Priming With Antigenically Mismatched Live Attenuated A/H7N3 Influenza Virus Vaccine Followed by Inactivated A/H7N9 Influenza Virus Vaccine
Brief Title: A Study in Healthy Adults to Assess Priming With Antigenically Mismatched Live Attenuated A/H7N3 Influenza Virus Vaccine Followed by Inactivated A/H7N9 Influenza Virus Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 16-003
Record Dates: First submitted 2018-06-26; First posted 2018-07-10 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- H7N3 pLAIV + H7N9 pIIV (Experimental): Participants will receive H7N3 pLAIV on Days 0 and 28, followed by H7N9 pIIV on Day 84.
  Interventions: Biological: H7N3 pLAIV; Biological: H7N9 pIIV

INTERVENTIONS:
Biological: H7N3 pLAIV — Approximately 10^7.0 fluorescent focus units (FFUs) administered intranasally by an Accuspray device
  Other Names: Live attenuated A/H7N3 influenza virus vaccine
Biological: H7N9 pIIV — 30 micrograms administered by intramuscular (IM) injection
  Other Names: Inactivated A/H7N9 influenza virus vaccine

SUMMARY:
The purpose of this study is to assess priming with antigenically mismatched live attenuated A/H7N3 influenza virus vaccine followed by inactivated A/H7N9 influenza virus vaccine in healthy adults.

DETAILED DESCRIPTION:
This study will assess priming with antigenically mismatched live attenuated A/H7N3 influenza virus vaccine (H7N3 pLAIV) followed by inactivated A/H7N9 influenza virus vaccine (H7N9 pIIV) in healthy adults.

Participants will receive a dose of H7N3 pLAIV on Days 0 and 28, followed by a single dose of H7N9 pIIV on Day 84.

On Days -2 and 26, participants will be admitted to an inpatient clinic. They will receive the H7N3 pLAIV vaccine on Days 0 and 28. They will remain in the clinic for 9 days after receiving the vaccine and until they are no longer shedding vaccine virus. An additional study visit will occur on Day 56.

On Day 84, participants will receive the H7N9 pIIV vaccine. Additional study visits will occur on Days 87, 91, 98, 112, 140, and 180. Study visits may include physical examinations, nasal washes, and blood and urine collection. Participants will be contacted by phone on Day 264 for follow-up health monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and non-pregnant, non-breastfeeding females between 18 years and 49 years of age, inclusive. Children will not be recruited or enrolled in this study because they are not in the apparent risk group, for safety considerations, and because of the need for isolation.
* Are in good health, as determined by medical history and targeted physical examination to ensure any existing medical diagnoses or conditions (except those exclusionary) are stable. More information on this criterion can be found in the protocol.
* Agree to storage of blood specimens for future research.
* Available for the duration of the trial. Subjects must be willing and able to remain within the Isolation Unit for the specified duration of confinement.
* Provide written informed consent prior to initiation of any study procedures, including future use of specimens.
* Female subjects of child-bearing potential must agree to use effective birth control methods for the duration of the study (for example, pharmacologic contraceptives including oral, parenteral, and transcutaneous delivery; condoms with spermicide; diaphragm with spermicide; intrauterine device; abstinence from heterosexual intercourse, surgical sterilization). All female subjects will be considered being of child bearing potential except those who have undergone hysterectomy or tubal ligation and those in whom menopause occurred at least 1 year prior to the study.
* Agrees not to participate in another clinical trial with an investigational product for the entire duration of the study.
* Female subjects of childbearing potential must have a negative urine and serum pregnancy test within 24 hours (urine) to 48 hours (serum) prior to study vaccination.

Exclusion Criteria:

* Pregnancy as determined by a positive human choriogonadotropin (beta-HCG) test.
* Currently breastfeeding or planning to breastfeed or become pregnant at some point during the duration of the study.
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, electrocardiogram (EKG) and/or laboratory studies including urine testing. Alanine aminotransferase (ALT) levels greater than 2 times the upper normal limit will be exclusionary at baseline, prior to vaccination.
* Any current illness requiring daily medication other than the following: vitamins, birth control, anti-hypertensive medication, antihistamines, anti-depressant medication, cholesterol-lowering medication, treatment for gastroesophageal reflux disease, and thyroid medication unless approved by the principal investigator (PI).
* Behavioral or cognitive impairment or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and cooperate with the study protocol.
* Previous enrollment in an H7 vaccine trial or in any study of an avian influenza vaccine.
* Seropositive to the H7N3 or H7N9 influenza A virus (serum HAI titer greater than 1:8).
* Positive urine drug toxicology test indicating narcotic use/dependency.
* Have medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a subject participating in the trial or would render the subject unable to comply with the protocol.
* Have a history of severe reactions following previous immunization with licensed or unlicensed influenza virus vaccines.
* Have known hypersensitivity or allergy to eggs, egg or chicken protein, or other components of the study vaccine.
* Allergy to oseltamivir as determined by subject report.
* Current diagnosis of asthma or reactive airway disease (within the past 2 years).
* History of Guillain-Barré Syndrome.
* Positive enzyme-linked immunosorbent assay (ELISA) and confirmatory Western blot tests for human immunodeficiency virus-1 (HIV-1).
* Positive ELISA and confirmatory test (e.g., recombinant immunoblot assay) for hepatitis C virus (HCV).
* Positive hepatitis B virus surface antigen (HBsAg) by ELISA.
* Known immunodeficiency syndrome.
* Use of corticosteroids (excluding topical preparations) or immunosuppressive drugs within 30 days prior to vaccination.
* Receipt of a live vaccine within 4 weeks or a killed vaccine within 2 weeks prior to study vaccination.
* History of asplenia
* Use of anticancer chemotherapy or radiation therapy (cytotoxic) within 36 months prior to vaccination.
* Have known active neoplastic disease or a history of any hematologic malignancy.
* Receipt of blood or blood-derived products (including immunoglobulin) within 6 months prior to study vaccination.
* Current smoker unwilling to stop smoking for the duration of the inpatient stay.

  * A current smoker includes anyone stating they currently smoke or use any amount of a tobacco product, including electronic cigarettes.
  * After admission to the unit, nicotine patches will be provided to current smokers who request them for the inpatient portion of the study.
* Travel to the Southern Hemisphere within 14 days prior to study vaccination.
* Travel on a cruise ship within 14 days prior to study vaccination.
* Receipt of another investigational vaccine or drug within 30 days prior to study vaccination.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2019-02-06 (Actual)

PRIMARY OUTCOMES:
Hemagglutination-inhibition (HAI) antibody response to H7N9 virus following administration of pIIV | Measured through Day 28
  Defined as 4-fold or greater response to a titer of 1:40 or above with 95% confidence intervals for both antigens

SECONDARY OUTCOMES:
Frequency of reactogenicity events following each dose of vaccine | Measured through Day 180
  Reactogenicity events will be collected and assessed for each individual subject, taking the pattern of viral shedding into account.
Severity of reactogenicity events following each dose of vaccine | Measured through Day 180
  Assessed according to the Reactogenicity Event Severity Grading System provided in the protocol
Frequency of adverse events following each dose of vaccine | Measured through Day 180
  All adverse events will be recorded and relationship to study product will be assessed.
Severity of adverse events following each dose of vaccine | Measured through Day 180
  Assessed according to the Adverse Event Severity Grading System provided in the study protocol
Frequency of vaccine viral shedding after each dose | Measured through Day 180
  Determined by rtRT-PCR and culture at each day tested after inoculation
Serum HAI and neutralizing antibody response following 1 or 2 doses of pLAIV | Measured through Day 56
  Response rates defined as 4-fold or greater response to a titer of 1:40 or above with 95% confidence intervals for both antigens
Neutralizing and HAI responses after pIIV boost against antigenic variants of H7 virus, including H7N7, H7N3, and H7N9 North American and Eurasian lineage viruses | Measured through Day 28
  Response rates defined as 4-fold or greater response to a titer of 1:40 or above with 95% confidence intervals for both antigens

CONTACTS AND LOCATIONS:
Overall Officials: Angela Branche, M.D., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center Vaccine Research Unit (Outpatient), Rochester, New York, United States